CLINICAL TRIAL: NCT04640272
Title: A Multi-Center, Open Label, TOFU Extension Study Assessing the Efficacy and Safety of Additional Intravitreal Injections of RBM-007 in Subjects With Wet Age-related Macular Degeneration
Brief Title: A Multi-Center, Open Label, Extension Study Assessing the Efficacy and Safety of Additional Intravitreal Injections of RBM-007 in Subjects With Wet Age-related Macular Degeneration
Acronym: RAMEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ribomic USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBM 007-003
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Exudative Age-related Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Open-label, non-comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RBM-007 injectable solution (Experimental): intravitreal injection
  Interventions: Drug: RBM-007

INTERVENTIONS:
Drug: RBM-007 — Intravitreal injection

SUMMARY:
This is a multi-center, open label, extension study of NCT04200248 assessing the efficacy and safety of additional intravitreal injections of RBM-007 in subjects with wet age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved Informed Consent Form (ICF) and provide authorization as appropriate for local privacy regulations.
2. Male or female 55 years of age or older on the date of signing the ICF and able and willing to comply with all treatment and study procedures.
3. Subjects must have completed all scheduled visits of previous study. Subjects can only enter this study after exiting previous study
4. Subjects for which previous previous masked treatment arms with intravitreal anti-vascular endothelial growth factor (anti-VEGF) agents Eylea® and/or RBM-007 has not demonstrated improvement in vision; subjects with less than 15 letter Best Corrected Visual Acuity (BCVA) improvement in TOFU study at exit visit over its baseline.
5. Diagnosis of exudative age-related macular degeneration (AMD) in the study eye, as assessed by spectral domain optical coherence tomography (SD-OCT).
6. Absence of central atrophy or retinal epithelial tear in the fovea or any condition preventing VA improvement in the study eye.
7. BCVA of 24 ETDRS letters (20/320) or better in the fellow eye.
8. Reasonably clear media and some fixation in the study eye to allow for good quality SD-OCT and fundus photography.

Exclusion Criteria:

* 1. Subjects whose vision have improved >15 BCVA letters at exit visit of previous study over its baseline 2. Subjects who experienced any drug related serious adverse event during previous study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Padma Bezwada, PhD, Study Director — Ribomic USA Inc
Locations (6):
- United States (6):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retinal Medical Consultants Group, Sacramento, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RBM-007 Injectable Solution
Started | 22
Completed | 21
Not Completed | 1
Not completed — Subject moved out of area | 1

BASELINE CHARACTERISTICS:
Arm/Group | RBM-007 Injectable Solution
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.41 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Best corrected visual acuity [Mean (Standard Deviation); unit: Letters seen on eye chart] | 61.82 (14.47)
Central macular subfield thickness [Mean (Standard Deviation); unit: microns] | 438.64 (129.69)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity - Continuous
Description: Mean change in Best Corrected Visual Acuity from Baseline
Time Frame: Month 4
Measure: Mean (Standard Deviation); unit: Letter seen on eye chart
Arm/Group | RBM-007 Injectable Solution
Number analyzed (Participants) | 22
Letter seen on eye chart | -5.5 (1.2)

2. Secondary Outcome: Visual Acuity - Categorical
Description: Percentage of patients gaining more than 15 letters as measured by Best Corrected Visual Acuity from Baseline
Time Frame: Month 4
Measure: Count of Participants; unit: Participants
Arm/Group | RBM-007 Injectable Solution
Number analyzed (Participants) | 22
Participants | 0

3. Secondary Outcome: Change From Baseline in Central Macular Subfield Thickness
Time Frame: Month 4
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | RBM-007 Injectable Solution
Number analyzed (Participants) | 22
Microns | 55.9 (15.66)

ADVERSE EVENTS:
Time Frame: Baseline through Month 4
Arm/Group | RBM-007 Injectable Solution
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBM-007 Injectable Solution (N=22)
COVID-19 (Infections and infestations) | 1 (1) — COVID-19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBM-007 Injectable Solution (N=22)
Infections and infestations (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04640272/Prot_000.pdf